CLINICAL TRIAL: NCT06963515
Title: Cutting-edge IMAGING Technologies to Improve the SAFEty and the Sustainability of LUNG Cancer Screening and the Accuracy of Non-invasive Lung Nodules Characterization
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Antonio Esposito, Professor, IRCCS San Raffaele
Other Study IDs: IMAGING-SAFE-LUNG
Record Dates: First submitted 2025-02-19; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer
Keywords: Magnetic Resonance Imaging; Low Dose Computed Tomography
MeSH Terms: conditions — Lung Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — 3T Magnetic Resonance Imaging

SUMMARY:
Low-dose computed tomography (LDCT) is used in individuals at high risk of developing lung cancer (smokers over 50 years of age), as it allows for the identification of pulmonary nodules, which, in a small percentage of cases, may represent early-stage lung cancer. However, according to LUNG-RADS guidelines, individuals undergoing screening must repeat multiple LDCT scans, as the comparison between successive LDCT scans enables the assessment of existing nodules' progression and the identification of newly developed pulmonary nodules. This results in cumulative exposure to ionizing radiation, increasing the risk of radiation-induced cancers.

This study addresses, through the implementation of new imaging techniques utilizing the latest and most advanced technological innovation (high-field 3T Magnetic Resonance Imaging (MRI) with artificial intelligence), the critical challenge of reducing radiation exposure in current LDCT-based screening programs, proposing the use of MRI as an alternative screening method to LDCT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Indication to first lung cancer screening with LDCT according to international guidelines
* Indication to repeated lung cancer screening with LDCT according to international guidelines

Exclusion Criteria:

* Age < 18 years
* contraindication to MRI
* presence of metallic implants likely to hamper MRI image quality
* inability to hold breath for 15-20 seconds
* claustrophobia
* refusal to participate in the study

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population will include 250 participants at high risk of lung cancer (smokers over 50 years old) already enrolled in screening programmes undergoing baseline or repeated CT scans.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2027-06-20 (Estimated); Study Completion 2028-06-20 (Estimated)

PRIMARY OUTCOMES:
the sensitivity and specificity for lung nodule detection of a Single Breath- Hold Lung non-contrast MRI scan (SBH-Lung-MRI), lasting less than 20 seconds, in comparison to LDCT | 3 years

SECONDARY OUTCOMES:
the sensitivity and specificity for lung nodule detection of SBH-Lung-MRI, lasting less than 20 seconds, in comparison to two of the most accurate available sequences for MRI lung nodule detection, namely: 2D-UTE and spiral 3D- UTE MRI sequences. | 3 years

OTHER OUTCOMES:
The health impact of implementing a radiation-free MRI-based lung cancer screening program using the SBH-Lung-MRI approach compared to conventional LDCT screening. | 3 years
  The following will be used to assess this outcome measures: number of lung cancer cases detected, stage distribution at detection, lung cancer-specific mortality, and overall mortality.
The cost-effectiveness of implementing a radiation-free MRI-based lung cancer screening program using the SBH-Lung-MRI approach tested in specific aim 1 compared to conventional LDCT screening. | 3 years
  The following will be used to assess this outcome measures: total program costs, costs per scan, and scanner operational efficiency (e.g., cost per hour of scanner use).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] de Koning HJ, van der Aalst CM, de Jong PA, Scholten ET, Nackaerts K, Heuvelmans MA, Lammers JJ, Weenink C, Yousaf-Khan U, Horeweg N, van 't Westeinde S, Prokop M, Mali WP, Mohamed Hoesein FAA, van Ooijen PMA, Aerts JGJV, den Bakker MA, Thunnissen E, Verschakelen J, Vliegenthart R, Walter JE, Ten Haaf K, Groen HJM, Oudkerk M. Reduced Lung-Cancer Mortality with Volume CT Screening in a Randomized Trial. N Engl J Med. 2020 Feb 6;382(6):503-513. doi: 10.1056/NEJMoa1911793. Epub 2020 Jan 29. PMID 31995683
- [Background] Potter AL, Rosenstein AL, Kiang MV, Shah SA, Gaissert HA, Chang DC, Fintelmann FJ, Yang CJ. Association of computed tomography screening with lung cancer stage shift and survival in the United States: quasi-experimental study. BMJ. 2022 Mar 30;376:e069008. doi: 10.1136/bmj-2021-069008. PMID 35354556
- [Background] Christensen J, Prosper AE, Wu CC, Chung J, Lee E, Elicker B, Hunsaker AR, Petranovic M, Sandler KL, Stiles B, Mazzone P, Yankelevitz D, Aberle D, Chiles C, Kazerooni E. ACR Lung-RADS v2022: Assessment Categories and Management Recommendations. J Am Coll Radiol. 2024 Mar;21(3):473-488. doi: 10.1016/j.jacr.2023.09.009. Epub 2023 Oct 10. PMID 37820837
- [Background] McCunney RJ, Li J. Radiation risks in lung cancer screening programs: a comparison with nuclear industry workers and atomic bomb survivors. Chest. 2014 Mar 1;145(3):618-24. doi: 10.1378/chest.13-1420. PMID 24590022
- [Background] Ohno Y, Takenaka D, Yoshikawa T, Yui M, Koyama H, Yamamoto K, Hamabuchi N, Shigemura C, Watanabe A, Ueda T, Ikeda H, Hattori H, Murayama K, Toyama H. Efficacy of Ultrashort Echo Time Pulmonary MRI for Lung Nodule Detection and Lung-RADS Classification. Radiology. 2022 Mar;302(3):697-706. doi: 10.1148/radiol.211254. Epub 2021 Nov 30. PMID 34846203
- [Background] Sommer G, Tremper J, Koenigkam-Santos M, Delorme S, Becker N, Biederer J, Kauczor HU, Heussel CP, Schlemmer HP, Puderbach M. Lung nodule detection in a high-risk population: comparison of magnetic resonance imaging and low-dose computed tomography. Eur J Radiol. 2014 Mar;83(3):600-5. doi: 10.1016/j.ejrad.2013.11.012. Epub 2013 Dec 4. PMID 24364923
- [Background] Heuvelmans MA, Walter JE, Peters RB, Bock GH, Yousaf-Khan U, Aalst CMV, Groen HJM, Nackaerts K, Ooijen PMV, Koning HJ, Oudkerk M, Vliegenthart R. Relationship between nodule count and lung cancer probability in baseline CT lung cancer screening: The NELSON study. Lung Cancer. 2017 Nov;113:45-50. doi: 10.1016/j.lungcan.2017.08.023. Epub 2017 Sep 1. PMID 29110848
- [Background] McWilliams A, Tammemagi MC, Mayo JR, Roberts H, Liu G, Soghrati K, Yasufuku K, Martel S, Laberge F, Gingras M, Atkar-Khattra S, Berg CD, Evans K, Finley R, Yee J, English J, Nasute P, Goffin J, Puksa S, Stewart L, Tsai S, Johnston MR, Manos D, Nicholas G, Goss GD, Seely JM, Amjadi K, Tremblay A, Burrowes P, MacEachern P, Bhatia R, Tsao MS, Lam S. Probability of cancer in pulmonary nodules detected on first screening CT. N Engl J Med. 2013 Sep 5;369(10):910-9. doi: 10.1056/NEJMoa1214726. PMID 24004118